CLINICAL TRIAL: NCT02154880
Title: Translation Evaluation of Aging, Inflammation and HIV in Lung Function
Brief Title: Translation Evaluation of Aging, Inflammation and HIV in Lung Function (TEAL)
Acronym: TEAL
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alison Morris, Professor, University of Pittsburgh
Other Study IDs: 13050317; 1R01HL120398-01A0 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-06-03 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: HIV; COPD; Pulmonary Disease; Aging
Keywords: HIV; lung; aging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva, blood, bronchial wash
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HIV positive under 50yo: PFT's, lab work, 6MWT, questionnaires, at baseline 18months and 36 months.
  Interventions: Procedure: PFT; Procedure: lab work; Procedure: 6MWT
- HIV negative under 50 yo: PFT's, lab work, 6MWT, questionnaires, at baseline 18months and 36 months.
  Interventions: Procedure: PFT; Procedure: lab work; Procedure: 6MWT; Other: questionnaires
- HIV positive over 50yo: PFT's, lab work, 6MWT, questionnaires, at baseline 18months and 36 months.
  Interventions: Procedure: PFT; Procedure: lab work; Procedure: 6MWT; Other: questionnaires
- HIV negative over 50yo: PFT's, lab work, 6MWT, questionnaires, at baseline 18months and 36 months.
  Interventions: Procedure: PFT; Procedure: lab work; Procedure: 6MWT; Other: questionnaires

INTERVENTIONS:
Procedure: PFT — Lung function endpoints of FVC, FEV1, FEV1/FVC, and FEF25-75% will be measured with the flow-volume loop recorder on a NDD EasyOne Pro system before and after bronchodilator administration.
  Other Names: Spirometry
Procedure: lab work — The blood will be processed for serum, plasma, and PBMCS, and a portion stored to be used for future use. A hemoglobin and Carboxyhemoglobin will be done in order to calculate the DLCO.
  Other Names: blood work
Procedure: 6MWT — The six-minute walk tests are performed in a 100-foot segment of straight hallway marked at 1-foot intervals.
  Other Names: six minute walk test
Other: questionnaires — TEAL, MMRC and ST. George's Questionnaire will be administered. They are paper questionnaires that inquire about respiratory symptoms, quality of life, smoking history and other health issues
  Other Names: survey
  Groups: HIV negative over 50yo; HIV negative under 50 yo; HIV positive over 50yo

SUMMARY:
Hypothesis;Aging modifies the risk of pulmonary dysfunction in HIV+ individuals.

The study is a multicenter, prospective observational study of aging and pulmonary function in HIV. The investigator will determine the prevalence and risk factors for lung dysfunction as quantified by pulmonary function testing in both younger (<50 years) and older (≥50 years) HIV+ and HIV-uninfected controls. The investigator will build on existing cohorts and enrich enrollment for individuals over the age of 50 while adjusting for important co-variates such as ART, smoking history, co-infections, and illicit drug use. Evaluations will be scheduled at baseline, 18 months, and 36 months. Study visits will consist of blood draw, questionnaires, and pulmonary function testing.

DETAILED DESCRIPTION:
All clinical procedures will be performed by a registered nurse. Bronchoscopy procedures will be performed by physician.

Subjects will be instructed to avoid smoking, alcoholic beverages and caffeine or medications containing caffeine for eight hours, prior to the visit. In addition, the subject will be asked to hold all medications that are bronchodilators prior to the test being administered and to eat a light meal 2-4 hours prior to testing.

Part I

Respiratory questionnaires:

Translation Evaluation of Aging, Inflammation and HIV in Lung Function questionnaire, MMRC and the ST. George's Questionnaire will be administered. These are paper and pencil questionnaires that inquire about respiratory symptoms, quality of life, smoking history and other health issures. This will take approximately 30 minutes to complete.

Blood Sample collection:

The subject will be asked to provide a blood sample by venipuncture of approximately 40mls (8 teaspoons) at this study visit. The purpose of this collection is to have blood processed for serum, plasma, and PBMCS, and a protion stored in RNAlater to be used for future use. A hemoglobin and Carboxyhemoglobin will be done in order to calculate the DLCO. The de-identified samples will be processed and stored at -80C.

Personal genetic information will not be provided to individual research subjects as Dr. Morris's laboratory is not CLIA certified and because the blood samples will be de-identified.

Lung function testing:

The routine lung function endpoints of FVC, FEV1, FEV1/FVC, and FEF25-75% will be measured with the flow-volume loop recorder on a NDD EasyOne Pro testing system before and after bronchodilator administration. The system is calibrated for body temperature and pressure of saturated gas and volumes, per American Thoracic Society (ATS) standards . The best of three reproducible forced expiratory attempts is used in analysis. Percent predicted spirometric values are based on age, height, gender, and ethnicity. DLco will be measured using the automated single-breath procedure of the integrated testing system, which conforms with ATS standards. All testing will be reviewed by (PI). If any concerns or abnormal results are discovered during this testing, a member of the research team will notify the subject or the subject's primary care physician, who will assess the need to provide additional evaluation.

Subjects will have these tests done at baseline, 18 months and 36 months. Each visit will last 3 to 4 hours. The visits will take place in the MUH 6th floor CTRC

6 minute walk test; Particiapant will rest for 10 minutes prior to beginning the test. BP and pulse ox are checked prior to the test. The six-minute walk tests are performed in a 100-foot segment of straight hallway marked at 1-foot intervals. In addition to the usual ATS protocol, the patient is monitored with wireless pulse oximetry and the time and distance recorded at which they desaturate to <88% or at 6 minutes. The test is also terminated if the saturation falls below 80%. Dyspnea and perceived exertion are rated using the Borg scale at the end of test. BP is checked post test. For this study the test will be performed off of supplemental oxygen if possible. O2 can be used on subjects who use O2 regularly to keep O2Sat > 88%

Oral specimen collection. The investigator will collect a 10ml oral wash, a tongue scraping and a 1 to 5ml saliva collection. This is a one time collection at any visit.

Part II Bronchoscopy visit (Selected subjects only) Subjects will be called back depending on the outcome of the PFT's and medical history. Subjects selected for bronchoscopy may have lung testing repeated depending on the time lapse between PFT and bronchoscopy. This will be decided at the discreation of the PI There will be two visits for the bronchoscopy participants. Both visits will take place in MUH 6th floor CTRC

Visit One: Apprx. 3 hours Screening procedures Oral Wash Tongue scraping Sputum induction Blood collection (Repeat breathing test will be completed at the discretion of the principal investigator)

Oral Wash The participant will gargle with .9% saline for 1 minute and then spit into a container to provide a sample of approximately 10mls (2 teaspoons) at this study visit.

Tongue Scraping A tongue blade or similar object will be used to scrape the tongue. This procedure should only take minutes.

Sputum Induction The subject will breathe in and out mists of saline (3%-5% saline) with a mouthpiece for 20 minutes. During this time, they will actively cough and spit out saliva and sputum into two separate cups every 4 minutes. We will frequently measure lung function during the procedure (every 4 min) using a peak flow meter.

Blood The investigator will take a blood sample of approximately 60mls (10 teaspoons) at this study visit for research blood. (serum, plasma, and PBMCS ) In addition, part of this blood will be used to perform routine clinical blood tests to assure that it is safe to proceed with the bronchoscopy test. (CBC/DIFF/PLT, LYTS, BUN, Creatinine, Glucose, PT/PTT)

Visit Two: Approx. 6 hours Oral wash Tongue scraping with rinse Bronchoscopy Monitoring (Blood draw- if visit two is more than 24 hours from visit one to repeat clinical labs)

Oral wash and Tongue Scraping will be repeated, and then the subject will rinse with 10cc's of Listerine. to assure that there are no bacteria left behind in the mouth prior to the bronchoscopy.

Bronchoscopy: Fiberoptic bronchoscopy will be performed using the ATS recommendation and institutional protocols for conscious sedation. The testing will be performed by a physician certified in pulmonary medicine and proficient in the procedure and certified by UPMC. Subjects will be instructed to fast overnight and withhold aspirin and anti-inflammatory analgesics for 48 hours prior to the procedure. Subjects will have undergone a pre- bronchoscopy spirometry and only clinically stable subjects (FEV1>30% predicted after albuterol) will undergo the procedure. Subjects will also recieve Proventil HFA Inhaler 2 puffs, after 5 minutes will recieve a second dose of Proventil 2 puffs prior to sending patient to the Bronchoscopy suite. Subjects will recieve an intramuscular injection of a mild sedative and a drug to dry secretions Demerol 50mg IV and Atropine 0.6mg.

Subjects will receive a local anesthetic to the upper and lower airways and an intravenous sedative and/or analgesic (midazolam; fentanyl). The midazolam dose will not exceed 10mg and/or the fentanyl dose will not exceed 200 micrograms. Lidocaine will not exceed a dose of 9 mg/kg (0.9 cc of 1%/kg) or a maximum dose of 600 mg (60 cc 1%) during the procedure. Subject monitoring will follow the local protocol for conscious/deep sedation. If needed, subjects will receive additional short acting beta agonist. After transoral insertion of the bronchoscope a general inspection of the airways will be performed followed by the bronchoalveolar lavage. Blood pressure, heart rate, and oxygen saturation will be monitored throughout the procedure.

Bronchoalveolar lavage:

BAL will be performed with room temperature normal saline. After wedging the bronchoscope in a (sub)segmental bronchus, approximately 50cc of saline will be instilled with each washing and withdrawn by syringe aspiration. This will be repeated up to 4 times per segment as needed. Amount of wash and selection of segments will be at the discretion of the physician. Many clinical bronchoscopies are within this range of volume, and research bronchoscopies have been found to be safe with volumes ranging from 100 to 300 cc even in subjects with severe asthma (Wenzel S et al. Bronchoscopic evaluation of severe asthma. American Journal of Respiratory and Critical Care Medicine 1997;156:737-43; Summary and recommendations of a workshop on the investigative use of fiberoptic bronchoscopy and bronchoalveolar lavage in asthmatic patients. Chest 1985;88:136-38). We will stop the lavage at any point where we do not feel that it would be clinically tolerated by the patient.

The volume collected after each withdrawal will be recorded.

Bronchial brushing:

Cytology bronchial brushing involves positioning the bronchoscope at the right middle or lower lobe, passing a cytology brush through the bronchoscope and gently brushing the lining of the airways. This may be repeated at least eight more times per segment to ensure an adequate sample collection. If any sample collected is not acceptable or adequate for analysis, another sample may be collected so long as the physician performnig the bronchoscopy procedure decides that no significant risk is present with the additional collection.

1. Participant will be monitored at UPMC Montefiore until the sedation has worn off. After the bronchoscopy is completed, the subject will wait in the bronchoscopy recovery area or the clinical research CTRC to make sure thier breathing has not been affected by the procedure and to be sure that the anesthesia has worn off. Pulse oximetry montioring will continue throughout recovery period. If the subject is not able to breathe as well as they could before the bronchoscopy, we will give additional albuterol and check the breathing again.Participant will not be allowed to leave the recovery area until their breathing is back to their normal level. If a participants breathing does not return to baseline they will be required to be admitted overnight
2. Participant will not be allowed to drive themselves home after the bronchoscopy.

Broncoscopy pre and post sedation care will be conducted in the MUH CTRC. Staff are trained research registered nurses and familiar with post bronchoscopy monitoring. Pulse oximetry will be closely monitored and the subect will not be discharged until anethseia has worn off and the subject's breathing is back to normal.

The bronchoscopy procedure will take about 45 minutes, the participant will not be discharged until anesthesia has worn off and their breathing is back to normal.

All bronchoscopies will be done in the pulmonary division bronchoscopy suite. Resuscitative equipment and personnel are present in the room to minimize risk. In addition, all research bronchoscopies will have an RN present, as well as the physician in charge of the procedure. The physician will be a faculty member of UPMC with brochoscopy privileges.

Bronchoscopy will only be offered once.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy or breast-feeding.
* Contraindication to pulmonary function testing (i.e. abdominal or cataract surgery within 3 months, recent myocardial infarction, etc.).
* Increasing respiratory symptoms or febrile (temperature >100.40F [380C]) within 4 weeks of study entry.
* Hospitalization within 4 weeks prior to study entry.
* Uncontrolled hypertension at screening visit (systolic > 160 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings. Subject may return for screening after blood pressure is controlled.
* Active cancer requiring systemic chemotherapy or radiation.
* Active infection of lungs, brain, or abdomen.
* Intravenous drug use or alcohol use that will impair ability to complete study investigations in the opinion of the investigator.

Exclusion Criteria:

HIV+ young:

* HIV-1 infection, documented in medical record at any time prior to study entry.
* Men and women age 45 years and below.
* Ability and willingness to complete all tests.
* Participant in MACS, Women's Interagency Health Study and secondarily clinics and the community

HIV+ old:

* HIV-1 infection, documented in medical record at any time prior to study entry.
* Men and women age 50 years and above.
* Ability and willingness to complete all tests.
* Participant in MACS, Women's Interagency Health Study and secondarily clinics and the community

HIV- young:

* HIV-uninfected, documented at most recent MACS or WIHS visit.
* Men and women age 45 years and below.
* Ability and willingness to complete all tests.
* Participant in MACS, Women's Interagency Health Study and secondarily clinics and the community

HIV- old:

* HIV-uninfected, documented at most recent MACS or WIHS visit.
* Men and women age 50 years and above.
* Ability and willingness to complete all tests.
* Participant in MACS, Women's Interagency Health Study and secondarily clinics and the community

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be subjects in the Pitt Men's Study or the PACT clinic.
Sampling Method: Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Number of HIV+ individuals with increased lung dysfunction disproportionate to age. | 2 years
  determine the prevalence and risk factors for lung dysfunction as quantified by pulmonary function testing in both younger (<50 years) and older (≥50 years) HIV+ and HIV-uninfected controls. We will build on existing cohorts and enrich enrollment for individuals over the age of 50 while adjusting for important co-variates such as ART, smoking history, co-infections, and illicit drug use.
Number of HIV COPD patients with increased immune cell and lung cellular aging. | 3 yrs
  We will attempt to proved the hypothesis that immune cell and lung cellular aging are increased in HIV COPD.We will examine telomere length and senescence markers in peripheral immune cells, lung immune cells and in lung epithelial cells and will test the hypothesis that HIV+ individuals with worse lung function and faster pulmonary decline manifest a greater degree of immune activation and cellular senescence.
Measurement of the inflammome in HIV-associated lung disease. | 4 years
  We will use this cohort to evaluate biomarkers of inflammation such as IL-6, IL-8, TNF-alpha, and hsCRP to determine if we can identify specific HIV COPD phenotypes using novel decision tree analyses. We will examine relationship of the inflammatory signature associated with COPD to aging markers in Aim 2, as well as ART effects, co-infections, degree of immunosuppression, and other co-variates.

SECONDARY OUTCOMES:
Measurement of Pulmonary immune cell senescence in HIV+ individuals with poor lung function. | 4 years
  we will test the hypothesis that HIV+ individuals with worse lung function and faster decline manifest a greater degree of pulmonary immune cell senescence and higher levels of senescence-associated cytokines.We will recruit a subset of 30 individuals and perform bronchoscopy with bronchoalveolar lavage (BAL). We will examine telomere length in alveolar macrophages (the primary cell obtained at BAL) and perform flow cytometry for markers of immune activation and senescence as in Aim 2a. We will also measure selected BAL cytokines (Table 2). Bronchoscopies will be performed only at the University of Pittsburgh site due to the need for immediate analyses and cell cultures.
The number of lung epithelial cell senescence in HIV+ individuals. | 4 years
  Bronchial epithelial cells are the most easily accessible lung cells, and these cells are likely to be important in the development of HIV COPD. The bronchial epithelium is an active part of the immune response and secretes chemoattractants and pro-inflammatory cytokines as well as matrix metalloproteases that could further perpetuate lung damage. The inflammation, injury, and repair cycle may lead to repeated cell turnover resulting in cellular senescence, apoptosis, and COPD. Lung epithelial cells in HIV- COPD patients display increased senescent markers including decreased telomere length18,19,26-28, but similar changes have not been investigated in HIV COPD. As part of bronchoscopy, we will collect human bronchial epithelial (HBE) cells from endobronchial brushings. Telomere length will be measured in HBE cells. These cells will also be cultured in air-liquid interface (ALI) and we will examine population doubling times, SA-ß-gal, and supernatant cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drummond MB, Huang L, Diaz PT, Kirk GD, Kleerup EC, Morris A, Rom W, Weiden MD, Zhao E, Thompson B, Crothers K. Factors associated with abnormal spirometry among HIV-infected individuals. AIDS. 2015 Aug 24;29(13):1691-700. doi: 10.1097/QAD.0000000000000750. PMID 26372280
- [Background] Qin S, Clausen E, Nouraie SM, Kingsley L, McMahon D, Kleerup E, Huang L, Ghedin E, Greenblatt RM, Morris A. Tropheryma whipplei colonization in HIV-infected individuals is not associated with lung function or inflammation. PLoS One. 2018 Oct 4;13(10):e0205065. doi: 10.1371/journal.pone.0205065. eCollection 2018. PMID 30286195
- [Background] Gingo MR, Nouraie M, Kessinger CJ, Greenblatt RM, Huang L, Kleerup EC, Kingsley L, McMahon DK, Morris A. Decreased Lung Function and All-Cause Mortality in HIV-infected Individuals. Ann Am Thorac Soc. 2018 Feb;15(2):192-199. doi: 10.1513/AnnalsATS.201606-492OC. PMID 29313714